CLINICAL TRIAL: NCT00806897
Title: Prospective, Multicentre, Open Label, Non-controlled, 24-week Observation in Type 2 Diabetics Using Once Daily Levemir® (Insulin Detemir) as Part of Their ITT Regimen
Brief Title: Observational Study in Type 2 Diabetics Treated by an Intensive Insulin Treatment of Levemir®
Acronym: LITHULEV1
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3701
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Effectiveness data collection in connection with the use of the drug Levemir® in daily clinical practice.
  Other Names: Levemir®; NN304

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to gain practical experience with once daily Levemir® administration in type 2 diabetes patients who were previously treated with NPH insulins (e.g. Protaphane®) as basal insulin as part of their IIT under normal clinical practice conditions in Lithuania

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic subjects on intensive insulin treatment (IIT)
* Eligibility for once daily insulin detemir administration
* Informed consent obtained before any observation-related activities

Exclusion Criteria:

* Known or suspected allergy to insulin detemir
* Subjects previously enrolled in the observation
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic subjects from specialists' (diabetologists, internists) care who are treated with intensive insulin treatment by prescription in line with governing prescribing rules. At baseline subjects are treated with IIT containing NPH as basal insulin.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | at 24 weeks

SECONDARY OUTCOMES:
Change in body weight | at 12 weeks/24weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Vilnius, Lithuania

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com